CLINICAL TRIAL: NCT04930094
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multicenter Phase III Trial to Investigate the Efficacy and Safety of Secukinumab 300 mg and 150 mg Administered Subcutaneously Versus Placebo, in Combination With a Glucocorticoid Taper Regimen, in Patients With Giant Cell Arteritis (GCA) (GCAptAIN)
Brief Title: Phase III Study of Efficacy and Safety of Secukinumab Versus Placebo, in Combination With Glucocorticoid Taper Regimen, in Patients With Giant Cell Arteritis (GCA)
Acronym: GCAptAIN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457R12301; 2024-510744-31-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: GCA; temporal arteritis; giant cell arteritis; vasculitis; secukinumab; monoclonal antibody; AIN457; prednisone taper regimen; glucocorticoid; GC
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 300 mg (Experimental): Secukinumab 300 mg s.c. at BSL, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4. Secukinumab will be given in combination with a specified 26-week prednisone taper regimen. After the 26-week prednisone taper, participants will continue to receive placebo to prednisone until Week 52.
  Interventions: Biological: Secukinumab 300 mg
- Placebo (Placebo Comparator): Placebo to secukinumab s.c. at BSL, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4. Placebo will be given in combination with a specified 52-week prednisone taper regimen.
  Interventions: Other: Placebo
- Secukinumab 150 mg (Experimental): Secukinumab 150 mg s.c. at BSL, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4. Secukinumab will be given in combination with a specified 26-week prednisone taper regimen. After the 26-week prednisone taper, participants will continue to receive placebo to prednisone until Week 52.
  Interventions: Biological: Secukinumab 150 mg

INTERVENTIONS:
Biological: Secukinumab 300 mg — Secukinumab 300 mg
  Other Names: AIN457
  Arms: Secukinumab 300 mg
Other: Placebo — Placebo
  Other Names: Placebo Comparator
  Arms: Placebo
Biological: Secukinumab 150 mg — Secukinumab
  Other Names: AIN457
  Arms: Secukinumab 150 mg

SUMMARY:
This is a phase III study of efficacy and safety of secukinumab versus placebo, in combination with glucocorticoid taper regimen, in patients with giant cell arteritis (GCA)

DETAILED DESCRIPTION:
Randomized, parallel-group, double-blind, placebo-controlled, multi-center, Phase III study to evaluate the efficacy and safety of secukinumab 300 mg and 150 mg administered subcutaneously versus placebo, in combination with a glucocorticoid taper regimen, in patients with giant cell arteritis (GCA) (GCAptAIN)

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study.
3. Male or non-pregnant, non-lactating female patients at least 50 years of age.
4. Diagnosis of GCA based on meeting all of the following criteria:

   * Age at onset of disease ≥ 50 years.
   * Unequivocal cranial symptoms of GCA (e.g., new-onset localized headache, scalp or temporal artery tenderness, permanent or temporary ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication), and/or unequivocal symptoms of polymyalgia rheumatica (PMR) (defined as shoulder and/or hip girdle pain associated with inflammatory morning stiffness) and/or symptoms of limb ischemia (claudication).
   * TAB revealing features of GCA and/or cross-sectional imaging study such as ultrasound (e.g., cranial or axillary), MRI/MRA, CTA, or PET-CT with evidence of vasculitis.
5. Active disease as defined by meeting both of the following within 6 weeks of BSL (see Section 8.1 for details)

   * Presence of signs or symptoms attributed to active GCA and not related to prior damage (e.g., visual loss that occurred prior to 6 weeks before BSL without new findings occurring within 6 weeks of BSL)
   * Elevated ESR ≥ 30 mm/hr or CRP ≥ 10 mg/L attributed to active GCA or active GCA on TAB or on imaging study.
6. Patients to meet definition of new-onset GCA or relapsing GCA:

   * Definition of new-onset GCA*: GCA that is diagnosed within 6 weeks of BSL visit
   * Definition relapsing GCA: GCA diagnosed > 6 weeks before BSL visit and following institution of an appropriate treatment course for GCA, participant has experienced recurrence of active symptoms or signs of disease after resolution.

     * The 6-week timeframe is to be calculated from the date of suspected GCA diagnosis. Suspected diagnosis is defined as date when GC therapy was initiated.
7. Patients' current GCA episode should be treatable with a dose of prednisone (or equivalent) designed to adequately achieve disease control in accordance with international guidelines. If this is not possible due to concerns regarding GC toxicity, the patient should not be enrolled. It must be medically appropriate for the patient to receive prednisone (or equivalent) 20 mg-60 mg daily (or equivalent) at BSL.
8. Patients taking MTX (≤ 25 mg/week) are allowed to continue their medication provided they have taken it for at least 2 months and are on a stable dose for at least 4 weeks prior to randomization and if they are on stable folic acid treatment before randomization.

Exclusion Criteria:

1. Pregnant or nursing (lactating) women where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
2. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during study treatment or longer if required by locally approved prescribing information (e.g., in European Union (EU) 20 weeks after treatment discontinuation). Also, contraception should be used in accordance with locally approved prescribing information of concomitant medications administered (e.g., Rescue Treatment). Effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Bilateral oophorectomy with or without hysterectomy, total hysterectomy or bilateral salpingectomy at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment are they not considered to be of child-bearing potential.
   * Bilateral tubal occlusion, Bilateral tubal ligation (at least six weeks before taking study treatment.
   * Male sterilization (vasectomy) of male partner(s) of the female participant at least 6 months prior to screening.
   * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps). NOTE: for United Kingdom: with spermicidal foam/gel/film/cream/vaginal suppository.
   * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS). In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
   * Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms). Women participants are considered not of child-bearing potential if they are post-menopausal or have had, surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral salpingectomy at least six weeks prior to first dose of study treatment in the study . In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered to be not of child-bearing potential.

   If local regulations are more stringent than the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the Informed Consent Form (ICF).
3. Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor.
4. Patients treated with any cell-depleting therapies.
5. Previous participation in a clinical trial where the outcome of treatment with the GCA drug is unknown. This does not include trials where the treatment for GCA was GCs, MTX, leflunomide or azathioprine
6. Patients who have been treated with inhibitors directly targeting IL-1, or IL-1 receptor, IL-12 and IL-23, or abatacept within 4 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL.
7. Treatment with tocilizumab, other IL-6/IL6-R inhibitor or JAK inhibitor within 12 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL, or if the patient did not respond to or experienced a relapse during treatment any time before BSL.
8. Any treatment received for GCA in which patient did not respond to treatment or experienced a relapse while on that treatment any time before BSL. This also includes patients who were treated in a clinical trial for GCA. Patients who failed on treatment with GCs, MTX, leflunomide and/or azathioprine may be included.
9. Patients treated with i.v. immunoglobulins or plasmapheresis within 8 weeks prior to BSL.
10. Patients treated (i.e. systemic therapy) with cyclophosphamide or hydroxychloroquine within 6 months prior to BSL, or tacrolimus, everolimus, cyclosporine A, azathioprine, sulfasalazine, mycophenolate mofetil within 4 weeks prior to BSL.
11. Patients treated with leflunomide within 8 weeks of BSL unless a cholestyramine washout has been performed in which case the patient must be treated within 4 weeks of BSL.
12. Patients treated with an alkylating agent within 5 years prior to BSL, unless specified in other exclusion criteria.
13. Patients requiring or anticipated to require systemic chronic glucocorticoid therapy or pulses of glucocorticoids for reasons other than GCA (e.g., COPD, asthma, planned surgery) at screening or randomization.
14. Criterion removed in protocol V01.
15. Patients requiring chronic (i.e., not occasional "prn") high potency opioid analgesics for pain management.
16. Use of other investigational drugs within 5 half-lives of enrollment or within 30 days (e.g. small molecules) or until the expected pharmacodynamic effect has returned to BSL (e.g., biologics), whichever is longer; or longer if required by local regulations.
17. History of hypersensitivity or contraindication to any of the study treatments or its excipients or to drugs of similar chemical classes.
18. Active IBD or other ongoing inflammatory diseases other than GCA that might confound the evaluation of the benefit of secukinumab therapy, including uveitis at screening or randomization.
19. Major ischemic event (e.g., myocardial infarction, stroke, etc.) or transient ischemic attack (TIA) (except ischemia-related vision loss), related or unrelated to GCA, within 12 weeks of screening.
20. Confirmed diagnosis of any primary form of systemic vasculitis, other than GCA.
21. Any other systemic biologics (e.g., denosumab, TNFα inhibitors) within 4 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL, or anticipated use of a systemic biologic prior to EOS
22. Active ongoing diseases which in the opinion of the investigator immunocompromises the patient and/or places the patient at unacceptable risk for treatment with immunomodulatory therapy.
23. Significant medical problems or diseases, including but not limited to the following: uncontrolled hypertension (≥ 160/95 mmHg), congestive heart failure (New York Heart Association (NYHA) status of class III or IV) and uncontrolled diabetes mellitus.
24. History of clinically significant liver disease or liver injury as indicated by abnormal liver function tests (LFTs) such as Aspartate Aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) or serum bilirubin. The investigator should be guided by the following criteria:

    * SGOT (AST) and SGPT (ALT) may not exceed 3 × the upper limit of normal (ULN). A single parameter elevated up to and including 3 × ULN should be re-checked once more as soon as possible, and in all cases, at least prior to randomization, to rule-out laboratory error.
    * Alkaline phosphatase may not exceed 2 × ULN. An elevation up to and including 2 × ULN should be re-checked once more as soon as possible, and in all cases, at least prior to randomization, to rule-out laboratory error.
    * Total bilirubin may not exceed 2 × ULN. If the total bilirubin concentration is increased above 2 × ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin.
25. Criterion removed in protocol V01
26. Screening total WBC count < 3,000/μL, or platelets < 100,000/μL or neutrophils < 1,500/μL or Hgb < 8.3 g/dL (83 g/L).
27. Active infections during the last 2 weeks prior to randomization.
28. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold Plus test. Patients with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active TB. If the test result is indeterminate, the investigator may repeat the test once or may proceed directly to perform the work-up for TB as per local procedures. If presence of latent TB is established then treatment according to local country guidelines must be initiated prior to randomization.
29. Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C (if not treated and cured) at screening or randomization
30. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
31. Live vaccinations (e.g., monkey pox vaccine, oral polio vaccine, varicella/zoster vaccines) within 6 weeks prior to BSL, or planned or anticipated potential need for live vaccination during study participation until 12 weeks after last study treatment administration.
32. Current severe progressive or uncontrolled disease, which in the judgment of the clinical investigator renders the patient unsuitable for the trial.
33. Any medical or psychiatric condition, which, in the investigator's opinion, would preclude the patient from adhering to the protocol or completing the study per protocol.
34. Donation or loss of 400 mL or more of blood within 8 weeks before randomization.
35. History or evidence of ongoing alcohol or drug abuse, within the last 6 months before randomization.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with sustained remission | 52 weeks
  Primary objective is to determine whether the efficacy of secukinumab 300 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week glucocorticoids (GC) taper regimen in participants with giant cell arteritis (GCA) based on sustained remission at Week 52

SECONDARY OUTCOMES:
Cumulative GC Dose | 52 weeks
  To demonstrate that the efficacy of secukinumab 300 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen, in participants with GCA, based on cumulative GC dose through Week 52
Proportion of participants with sustained remission | 52 weeks
  To demonstrate that the efficacy of secukinumab 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen in participants with GCA based on sustained remission at Week 52
Cumulative GC Dose | 52 Weeks
  To demonstrate that the efficacy of secukinumab 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen, in participants with GCA, based on cumulative GC dose through Week 52
Time to first use of Escape or Rescue Treatment due to GCA as measured in days | 52 weeks
  To demonstrate that the efficacy of secukinumab 300 mg s.c. or 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen in participants with GCA based on time to first use of Escape Treatment or Rescue Treatment due to GCA
Change in SF-36 score (PCS) | 52 weeks
  To demonstrate that the effect on participant's QoL of secukinumab 300 mg s.c. or 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen, in participants with GCA based on change of SF-36 score (PCS) at Week 52
Glucocorticoid Toxicity Index (GTI) as measured by the Aggregate Improvement Score (AIS) | 52 weeks
  To demonstrate that the effect of secukinumab 300 mg s.c. or 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen, in participants with GCA based on Glucocorticoid Toxicity Index (GTI)
Change in FACIT-Fatigue Score | 52 weeks
  To demonstrate that the effect on participant's QoL of secukinumab 300 mg s.c. or 150 mg s.c. in combination with a 26-week GC taper regimen is superior to placebo in combination with a 52-week GC taper regimen, in participants with GCA based on change in FACIT-Fatigue score at Week 52
Number of participants with Adverse events (AEs) and Serious AEs (SAEs) | 52 weeks
  Number of participants with AEs and SAEs as a measure of safety and tolerability
Number of participants with clinically significant changes in clinical laboratory measures and vital signs | 52 weeks
  Number of participants with clinically significant changes in clinical laboratory measures and vital signs, as assessed by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (99):
- United States (10):
  - Cedars Sinai Medical Center, Los Angeles, California
  - IRIS Research and Development, Plantation, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - Novartis Investigative Site, Iowa City, Iowa
  - University Of Iowa, Iowa City, Iowa
  - Osteoporosis and Clinical Trial Ctr, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - West Tennessee Research Institute, Jackson, Tennessee
  - Precision Comp Clin Research, Grapevine, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
- Argentina (2):
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Capital Federal
- Australia (7):
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Heidelberg Heights, Victoria
  - Novartis Investigative Site, Malvern East, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Parramatta
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
- Novartis Investigative Site, Plovdiv, Bulgaria
- Canada (3):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (3):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Vejle
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (4):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Lahti
  - Novartis Investigative Site, Turku
- France (9):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (9):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ludwigshafen
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Siena, SI
- Norway (2):
  - Novartis Investigative Site, Gjettum
  - Novartis Investigative Site, Moss
- Poland (2):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Malmo, Sweden
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
- United Kingdom (4):
  - Novartis Investigative Site, Edinburgh, Scotland
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Dundee

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com